CLINICAL TRIAL: NCT00945191
Title: Phase 2 Study of CS-1008 in Combination With Chemotherapy (Paclitaxel/Carboplatin) in Locally Advanced or Metastatic Ovarian Cancer
Brief Title: Combination Chemotherapy With CS-1008 to Treat Ovarian Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CS1008-A-U205
Record Dates: First submitted 2009-07-22; First posted 2009-07-24 (Estimated); Results first posted 2020-11-18 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-03

CONDITIONS: Ovarian Cancer Stage IIIC; Ovarian Cancer Stage IV
Keywords: Ovarian Cancer Stage IIIC; Ovarian Cancer Stage IV; CS-1008; Paclitaxel; Carboplatin
MeSH Terms: conditions — Ovarian Neoplasms | interventions — tigatuzumab; Paclitaxel; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CS-1008 with paclitaxel and carboplatin (Experimental): CS-1008 will be administered with paclitaxel and carboplatin.
  Interventions: Drug: CS-1008; Drug: Paclitaxel; Drug: Carboplatin

INTERVENTIONS:
Drug: CS-1008 — CS-1008 intravenous (IV) infusion 10 mg/kg on Day 1 of Cycle 1 and 8 mg/kg once every 3 weeks (1 cycle) for Cycle 2-6
Drug: Paclitaxel — Paclitaxel 175 mg/m^2 IV infusion once every 3 weeks (1 cycle) for 6 cycles
  Other Names: Taxol
Drug: Carboplatin — Carboplatin (target area under the concentration versus time curve of 6.0 mg/mL/min using the Calvert Formula) IV infusion once every 3 weeks (1 cycle) for 6 cycles

SUMMARY:
This trial assessed the effect of treatment with CS-1008 in combination with paclitaxel/carboplatin on response in patients with locally advanced or metastatic ovarian cancer.

DETAILED DESCRIPTION:
This trial assessed CS-1008 administered in combination with paclitaxel/carboplatin to patients with Stage IIIC or IV ovarian cancer who had suboptimal debulking surgery with residual measurable/evaluable disease and who had not received prior therapy for their disease. The effect of this first-line treatment in patients was assessed by complete response rate.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed, epithelial carcinoma of the ovary or primary peritoneal carcinoma (International Federation of Gynecology and Obstetrics [FIGO] Stage IIIC or IV).

(Participants with the following histologic epithelial cell types are eligible for the study: serous adenocarcinoma, endometrioid adenocarcinoma, mucinous adenocarcinoma, undifferentiated carcinoma, clear cell adenocarcinoma, mixed epithelial carcinoma, transitional cell carcinoma, malignant Brenner's Tumor, or adenocarcinoma not otherwise specified.)

* Enrollment within 6 weeks after surgical resection (debulking).
* Residual tumor masses > 1 cm and objectively measurable/evaluable disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST) criteria.
* No prior therapy for ovarian cancer (ie, chemotherapy or radiotherapy [RT] to the abdomen or pelvis) other than surgical debulking of disease.
* At least 18 years of age.
* Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 2.
* Adequate organ and bone marrow function as evidenced by:

  * Absolute neutrophil count ≥ 1,500/µL (equivalent to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), Version 3.0 grade 1)
  * Platelet count ≥ 100,000/µL (CTCAE grade 0 to 1)
  * Hemoglobin ≥ 9 g/dL
  * Serum creatinine ≤ 1.5 x institutional upper limit of normal (ULN) (CTCAE grade 1)
  * Bilirubin ≤ 1.5 x ULN (CTCAE grade 1)
  * Aspartate aminotransferase (AST) and alkaline phosphatase ≤ 2.5 x ULN (CTCAE grade 1)
* Adequate neurologic function (ie, sensory and motor neuropathy ≤ CTCAE grade 1).
* Women of childbearing potential must be willing to consent to using effective contraception while on treatment and for 3 months thereafter.
* All subjects of childbearing potential must have a negative pregnancy test (serum or urine) result ≤ 72 hours before initiating study treatment.
* Participants must be fully informed about their illness and the investigational nature of the study protocol (including foreseeable risks and possible side effects) and must sign and date an institutional review board-approved informed consent form (ICF) before performance of any study-specific procedures or tests.

Exclusion Criteria:

* Prior invasive malignant disease within 5 years except for squamous cell or basal cell carcinoma.
* Current diagnosis of borderline epithelial ovarian tumor (formerly "tumors of low malignant potential") or recurrent ovarian epithelial cancer.
* Positive human immunodeficiency virus (HIV) or hepatitis B surface antigen (HBsAg) because of the potential for additional toxicity from the treatment regimen.
* Anticipation of need for a major surgical procedure or radiotherapy (RT) during the study.
* History of any of the following conditions within 6 months before study enrollment: myocardial infarction; severe/unstable angina pectoris; coronary/peripheral artery bypass graft; New York Heart Association (NYHA) class III or IV congestive heart failure; cerebrovascular accident or transient ischemic attack, pulmonary embolism, or other clinically significant thromboembolic event; clinically significant pulmonary disease (eg, severe chronic obstructive pulmonary disease or asthma).
* Clinically active brain metastasis (ie, untreated, still requiring therapy with steroids or RT, or with progression within 4 weeks after completion of RT); an uncontrolled seizure disorder; spinal cord compression; or carcinomatous meningitis.
* Pregnant or lactating.
* Prior treatment with CS-1008, other agonistic DR5 antibodies, or tumor necrosis factor-related apoptosis inducing ligand (TRAIL).
* Known history of hypersensitivity reactions to any of the components of CS-1008, paclitaxel (or docetaxel), or carboplatin formulations.
* Serious intercurrent medical or psychiatric illnesses or any other conditions that in the opinion of the Investigator would impair the ability to give informed consent or unacceptably reduce protocol compliance or safety of the study treatment.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2009-10-06 (Actual); Primary Completion 2011-08-23 (Actual); Study Completion 2011-08-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Daiichi Sankyo
Locations (3):
- United States (3):
  - Univ. Alabama, Birmingham, Alabama
  - Barnes Jewish Hospital, St Louis, Missouri
  - University of Oklahoma, Oklahoma City, Oklahoma

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 24 participants who met all inclusion criteria and no exclusion criteria were enrolled and received treatment at 3 clinic sites in the United States.
Pre-assignment Details: Following debulking surgery, participants with suboptimal resection (ie, residual tumor > 1 cm) and measurable/evaluable tumor by imaging techniques were eligible for participation in this study. Debulking surgery occurred within 6 weeks before enrollment in the study.
Groups:
- CS-1008 in Combination With Paclitaxel/Carboplatin: Participants who received CS-1008 in combination with paclitaxel and carboplatin. CS-1008 was administered as an intravenous (IV) infusion 10 mg/kg on Day 1 of Cycle 1 and 8 mg/kg once every 3 weeks (1 cycle) for Cycle 2-6. Paclitaxel 175 mg/m^2 was administered as an IV infusion once every 3 weeks (1 cycle) for 6 cycles. Carboplatin (target area under the concentration versus time curve of 6.0 mg/mL/min using the Calvert Formula) was administered as an IV infusion once every 3 weeks (1 cycle) for 6 cycles.
Period: Overall Study
Arm/Group | CS-1008 in Combination With Paclitaxel/Carboplatin
Started | 24
Completed | 0
Not Completed | 24
Not completed — Did not achieve a complete response | 18
Not completed — Participant relocated to another state | 1
Not completed — Disease progression | 3
Not completed — Serious adverse event or adverse event | 1
Not completed — Investigator's discretion | 1

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were assessed in the Safety Analysis Set.
Arm/Group | CS-1008 in Combination With Paclitaxel/Carboplatin
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 17
  >=65 years | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.3 (9.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 22
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 24

OUTCOME MEASURES:

1. Primary Outcome: Best Overall Response and Objective Response Rate Following Treatment With CS-1008 in Combination With Chemotherapy (Paclitaxel/Carboplatin) in Locally Advanced or Metastatic Ovarian Cancer
Description: The best overall response is the best response (in the order of confirmed complete response [CR], confirmed partial response [PR], unconfirmed CR, unconfirmed PR, stable disease [SD], and progressive disease [PD]) among all overall responses recorded from the start of treatment until the participant withdraws from the study. If there is no tumor assessment after the first dose of study drug, the best overall response is classified as Inevaluable. CR was defined as a disappearance of all target lesions, PR was defined as at least a 30% decrease in the sum of diameters of target lesions, and SD was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD defined as at least a 20% increase in the sum of diameters of target lesions. Objective response rate was defined as confirmed CR and confirmed PR.
Time Frame: Baseline up to first documented objective response, disease progression, or study withdrawal, up to 1 year 10 months
Population: Best overall tumor response and objective response rate were assessed in the Full Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | CS-1008 in Combination With Paclitaxel/Carboplatin
Number analyzed (Participants) | 24
Participants
  Confirmed CR after 6 cycles (18 weeks) of treatment | 0
  Confirmed CR | 0
  Confirmed PR | 12
  Objective Response (Confirmed CR + Confirmed PR) | 12
  Unconfirmed CR | 0
  Unconfirmed PR | 4
  Stable disease (SD) | 5
  Progressive disease (PD) | 1
  Inevaluable | 2
  Best overall response of SD or better | 21

2. Secondary Outcome: Change From Baseline in the Sum of Longest Diameters of Target Lesions Following Treatment With CS-1008 in Combination With Chemotherapy (Paclitaxel/Carboplatin) in Locally Advanced or Metastatic Ovarian Cancer
Description: A sum of the diameters for all target lesions will be calculated and reported as the baseline sum of diameters, defined as the last non-missing value before initial administration of study treatment. The baseline sum of diameters will be used as reference for characterization of the objective tumor response. The change from baseline in the sum of longest diameters of target lesions is being reported. Negative values indicate an improvement in tumor reduction.
Time Frame: Baseline to Cycle 3, Week 3 Day 1; Cycle 6, Week 3 Day 1 (each cycle 21 days) up to end of study, approximately 1 year 10 months postdose
Population: The sum of longest diameters of target lesions was assessed in the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | CS-1008 in Combination With Paclitaxel/Carboplatin
Number analyzed (Participants) | 24
mm
  Cycle 3, Week 3 Day 1: number analyzed (Participants) | 21
  Cycle 3, Week 3 Day 1 | -39.0 (41.73)
  Cycle 6, Week 3 Day 1: number analyzed (Participants) | 19
  Cycle 6, Week 3 Day 1 | -52.4 (41.56)
  Minimum post-treatment value: number analyzed (Participants) | 21
  Minimum post-treatment value | -48.3 (41.65)

3. Secondary Outcome: Participants With Treatment-Emergent Adverse Events Grade 3 or Higher by System Organ Class and Preferred Term Following Treatment With CS-1008 in Combination With Chemotherapy (Paclitaxel/Carboplatin) in Locally Advanced or Metastatic Ovarian Cancer
Description: Treatment-emergent adverse events (TEAEs) were defined as those events that occur, having been absent before the study, or worsen in severity after the initiation of CS-1008 and/or paclitaxel/docetaxel/carboplatin administration. All adverse events (AEs) were graded (1 to 5) according to the National Cancer Institute Common Terminology Criteria for Adverse Events, Version 3.0, where Grade 1 was mild, Grade 2 moderate, Grade 3 severe, Grade 4 life-threatening or disabling, and Grade 5 death related to AE.
Time Frame: Baseline up to 30 days after last dose, up to 1 year 10 months postdose
Population: Treatment-emergent adverse events were assessed in the Safety Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | CS-1008 in Combination With Paclitaxel/Carboplatin
Number analyzed (Participants) | 24
Participants
  Any TEAE ≥Grade 3 | 22
  Any Preferred Term Within Blood and Lymphatic System Disorders | 20
  Anaemia | 6
  Febrile neutropenia | 1
  Leukopenia | 2
  Neutropenia | 18
  Pancytopenia | 1
  Thrombocytopenia | 7
  Any Preferred Term Within Gastrointestinal Disorders | 6
  Abdominal pain | 1
  Ascites | 2
  Constipation | 1
  Enterocolitis | 1
  Gastrooesophageal reflux disease | 1
  Small intestinal obstruction | 3
  Any Preferred Term Within General Disorders and Administration Site Conditions | 2
  Chills | 1
  Fatigue | 1
  Any Preferred Term Within Infections and Infestations | 3
  Abdominal abscess | 1
  Urinary tract infection | 3
  Wound infection staphylococcal | 1
  Any Preferred Term Within Investigations | 1
  Prothrombin time prolonged | 1
  Any Preferred Term Within Metabolism and Nutrition Disorders | 5
  Dehydration | 2
  Electrolyte imbalance | 1
  Hyperglycaemia | 1
  Hypokalaemia | 2
  Hyponatraemia | 1
  Hypophosphataemia | 1
  Any Preferred Term Within Musculoskeletal and Connective Tissue Disorders | 2
  Arthralgia | 1
  Back pain | 1
  Musculoskeletal pain | 1
  Any Preferred Term Within Renal and Urinary Disorders | 1
  Renal vein thrombosis | 1
  Any Preferred Term Within Vascular Disorders | 1
  Venous thrombosis | 1

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) were collected from baseline up to 30 days after last dose, up to 1 year 10 months postdose.
Description: Treatment-emergent adverse events (TEAEs) were defined as those events that occur, having been absent before the study, or worsen in severity after the initiation of CS-1008 and/or paclitaxel/docetaxel/carboplatin administration.
Arm/Group | CS-1008 in Combination With Paclitaxel/Carboplatin
All-Cause Mortality (participants affected / at risk) | 0/24
Serious Adverse Events (participants affected / at risk) | 9/24
Other Adverse Events (participants affected / at risk) | 11/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CS-1008 in Combination With Paclitaxel/Carboplatin (N=24)
Anaemia (Blood and lymphatic system disorders) | 3
Neutropenia (Blood and lymphatic system disorders) | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 2
Enterocolitis (Gastrointestinal disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 3
Abdominal abscess (Infections and infestations) | 1
Dehydration (Metabolism and nutrition disorders) | 2
Electrolyte imbalance (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Venous thrombosis (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CS-1008 in Combination With Paclitaxel/Carboplatin (N=24)
Anaemia (Blood and lymphatic system disorders) | 3
Neutropenia (Blood and lymphatic system disorders) | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Enterocolitis (Gastrointestinal disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 1
Abdominal abscess (Infections and infestations) | 1
Dehydration (Metabolism and nutrition disorders) | 2
Electrolyte imbalance (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Venous thrombosis (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No